CLINICAL TRIAL: NCT01364324
Title: Absorption of Anti-tuberculosis Drugs and Its Effect to Treatment Response in Gastrectomized Patients
Brief Title: Pharmacokinetics of Anti-tuberculosis Drugs in Gastrectomized Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Hee Seok Lee, Pulmonologist, National Cancer Center, Korea
Other Study IDs: NCCCTS-10-493
Record Dates: First submitted 2011-05-23; First posted 2011-06-02 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Early Gastric Cancer
Keywords: tuberculosis; pharmacokinetics; first-line drugs; gastrectomy
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastrectomy: Twenty gastrectomized patients with pulmonary TB, treated with standard first line anti-TB drugs(isoniazid/rifampicin/ethambutol/pyrazinamide), administered daily, orally
  Interventions: Drug: standard first line anti-TB drugs
- Non-gastrectomy: Twenty non-gastrectomized patients with pulmonary TB, treated with standard first line anti-TB drugs(isoniazid/rifampicin/ethambutol/pyrazinamide), administered daily, orally
  Interventions: Drug: standard first line anti-TB drugs

INTERVENTIONS:
Drug: standard first line anti-TB drugs — We will perform pharmacokinetic study in gastrectomy and non-gastrectomy group, to evaluate the effect of gastrectomy on pharmacokinetic profile of first-line anti-TB drugs in patients with TB
  Other Names: Pharmacokinetics of Anti-tuberculosis Drugs

SUMMARY:
The purpose of this study is to evaluate the effect of gastrectomy on pharmacokinetic profile of first-line anti-tuberculosis drugs in patients with pulmonary tuberculosis (TB).

DETAILED DESCRIPTION:
Gastrectomy is a well-known risk factor for TB. Also, there were some reports about malabsorption of anti-TB drugs in the gastrectomized patients. However, pharmacokinetics of recently used first line anti-TB drugs in the gastrectomized patients have not been well evaluated simultaneously. Therefore, the investigators aim to evaluate the effect of gastrectomy on pharmacokinetic profile of first-line anti-TB drugs in patients with pulmonary TB through this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years and less than 80 years
2. pulmonary TB confirmed by microbiologic test such as AFB culture or TB PCR
3. usage of 4 first-line anti-TB drugs (Isoniazid(INH) Rifampin(RFP) Ethambutol(EMB), Pyrazinamide(PZA) = HREZ)

Exclusion Criteria:

1. patients with liver disease (bilirubin ≥ 1.5 mg/d or AST ≥ 2 x normal upper limit) or chronic renal failure (Cr ≥ 2.0 mg/d) who cannot use first-line anti-TB drugs
2. patients with AIDS or hypoalbuminemia(albumin < 3.0g/dl)that will influence pharmacokinetics of first line anti-TB drugs
3. patients using other drugs that will influence pharmacokinetics of first line anti-TB drugs during anti-TB treatment (e.g warfarin)
4. patients using anti-cancer or immunosuppressive agents that will influence the response of pulmonary TB to anti-TB drugs
5. discontinuation of first-line anti-TB drugs(HREZ)due to side effect or resistance
6. follow-up loss before completion of anti-TB treatment
7. any condition making the patients undergo gastrectomy during anti-TB treatment in case of Non-gastrectomy group

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients with pulmonary TB diagnosed in our hospital and treated with 4 first line anti-TB drug(isoniazid/rifampicin/ethambutol/pyrazinamide= HREZ), we recruit patients who underwent gastrectomy to Gastrectomy group. And then, we recruit age-sex matched patients who did not underwent gastrectomy to Non-gastrectomy group.(age ±3 years)
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
The change in the maximum concentration (Cmax) of first-line TB drugs | Before and 1, 2, 4, 6 and 8 hours after dosing

SECONDARY OUTCOMES:
The effects of pharmacokinetics on responses of pulmonary TB to anti-TB drug | 9month after anti-TB treatment
  Treatment duration can be varied according to several factors such as a first TB episode or not, cavitary TB, and AFB culture(+) after 2month-treatment etc. We will plan 6 or 9 months treatment for each patient according to these factors. During treatment period, we will check chest radiographs and sputum AFB smear/culture with every 2-3month intervals. At 9month after treatment, we will evaluate the effects of pharmacokinetics on responses of pulmonary TB to anti-TB drug by taking account of improvement on chest radiograph and negative conversion and its continuation on sputum smear/culture.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seok Lee, M.D., Principal Investigator — National Cancer Center
Locations (1):
- Respiratory Clinic, National Cancer Center, Goyang-si, Gyeonggi-do, South Korea